CLINICAL TRIAL: NCT02089438
Title: Comparison of Three DPP-4 Inhibitors on 24 Hour Blood Glucose, Incretin Hormones and Islet Function in Patients With Type 2 Diabetes
Brief Title: DPP-4 Inhibition, Incretins and Islet Function
Acronym: CODI24
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200A
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Vildagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saxagliptin (Experimental): Ssaxagliptin is given before breakfast
  Interventions: Drug: Saxagliptin
- ´Sitagliptin (Experimental): Sitagliptin is given before breakfast
  Interventions: Drug: Sitagliptin
- Vildagliptin (Experimental): Vildagliptin is given before breakfast
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Saxagliptin — Saxagliptin (5 mg) is given before breakfast
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Vildagliptin — Vildagliptin (50mg) is given before breakfast and dinner
  Other Names: Galvus
  Arms: Vildagliptin
Drug: Sitagliptin — Sitagliptin (100 mg) is given before breakfast
  Other Names: Januvia
  Arms: ´Sitagliptin

SUMMARY:
Hypothesis is that DPP-4 inhibition affects glucose levels through changes in incretin and islet hormones. The study examines this in relation to breakfast, lunch and dinner over an entire 24h study period by the use of three different DPP-4 inhibitors and placebo.

DETAILED DESCRIPTION:
The study is a single-center study with a cross-over design to examine glycemia, incretin hormones and islet hormones over a 24h study period with standardized breakfast, lunch and dinner after administration of placebo, saxagliptin, vildagliptin or sitagliptin.

ELIGIBILITY:
Inclusion Criteria:

* • Caucasian men or women with type 2 diabetes diagnosed according to ICD10 at time of inclusion

  * Ongoing treatment with life style adjustment including diet and exercise regimen together with metformin as oral antidiabetic . Metformin therapy should be stable the last three months
  * Age 40-75 years
  * HbA1c 52-80 mmol/mol (inclusive)
  * BMI: 20-40 kg/m2
  * Written informed consent has been given
  * Capability and willingness to participate in the whole study

Exclusion Criteria:

* • Liver disease (K70-77 in ICD10) or liver enzymes three times above upper reference range

  * Diabetic nephropathy (GFR < 30 mL/min/1.73 m2 or albuminuria) or other causes of renal disease
  * Proliferative diabetic retinopathy
  * Treatment with any glucose-lowering medication except metformin
  * Previous myocardial infarction, coronary heart disease or instable angina pectoris in the last 6 months.
  * Symptomatic heart failure (NYHA class II-III)
  * Previous surgery on the gastrointestinal tract
  * Larger surgical intervention during the last 12 weeks
  * Female subject who are pregnant or breast feeding
  * Women of child bearing potential not using a highly effective method of birth control
  * Treatment with oral steroids, thiazide diuretics, digoxin or growth hormone
  * Hypersensitivity to the active substances of to any of the excipients
  * Participation in another study the last 4 weeks
  * Smoker
  * Paracetamol intolerance

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | 180 min
  The area under the 180 min curves for plasma glucose after each meal

SECONDARY OUTCOMES:
Postprandial insulin and glucagon | 180 min
  The area under the 180 min curves for plasma insulin and glucagon after each meal
Postprandial glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) | 180 min
  The area under the 180 min curves for plasma GLP-1 and GIP after each meal

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Clinical Research Department, Lund, Sweden